CLINICAL TRIAL: NCT05635890
Title: Effect of Vestibular Rehabilitation on Trunk Kinetic and Kinematic Parameters in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Ahmed Magdy Alshimy, Lecturer of Physical Therapy at department of neurology, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003988
Record Dates: First submitted 2022-11-13; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Vestibular Rehabilitation in MS
Keywords: Trunk kinetic and kinematic parameters, Vestibular rehabilitation, Multiple Sclerosis.
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): received conventional vestibular rehabilitation along with the Cawthorne Cooksey exercise protocol
  Interventions: Other: Cawthorne Cooksey exercise protocol; Other: conventional vestibular rehabilitation
- Group II (Active Comparator): received conventional vestibular rehabilitation only
  Interventions: Other: conventional vestibular rehabilitation

INTERVENTIONS:
Other: Cawthorne Cooksey exercise protocol — Cawthorne Cooksey exercise protocol
  Arms: Group I
Other: conventional vestibular rehabilitation — conventional vestibular rehabilitation

SUMMARY:
The Cawthorne Cooksey exercises and conventional program of physical therapy were administered.

DETAILED DESCRIPTION:
• The Cawthorne Cooksey exercises and conventional program of physical therapy were administered.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-55 years.
* Ambulatory without assistance.
* Diagnosed with relapsing-remitting MS by a neurologist, with approximately five relapse attacks in the hemiparesis type with a muscular tone of 1 or 1+ depending on the MAS, or modified Ashworth scale.
* All individuals were evaluated by a neurosurgeon to confirm central vertigo using test of Dix Hallpike.
* Degree of MS-related disability based on the enlarged disability status scale, ranging from 2-2.5.

Exclusion Criteria:

* People with musculoskeletal deformities.
* People with inner ear abnormalities.
* People with psychiatric disturbances or seizures.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Isokinetic dynamometer (average power) | 4 weeks
  Assess trunk kinetic and kinematic parameters.
Isokinetic dynamometer (acceleration time) | 4 weeks
  Assess trunk kinetic and kinematic parameters.
Isokinetic dynamometer (deceleration time) | 4 weeks
  Assess trunk kinetic and kinematic parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No